CLINICAL TRIAL: NCT02022306
Title: A Double-Blinded, Randomized, Placebo-Controlled, Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Food Effect of TD-6450, a NS5A Inhibitor, in Healthy Subjects
Brief Title: TD-6450 SAD and MAD in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0094
Record Dates: First submitted 2013-12-17; First posted 2013-12-27 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- SAD TD-6450 (Placebo Comparator): Single ascending dose (Part A)
  Interventions: Drug: TD-6450; Drug: Placebo
- MAD TD-6450 (Placebo Comparator): Multiple ascending dose (Part B)
  Interventions: Drug: TD-6450; Drug: Placebo
- Food effect of TD-6450 (Active Comparator): Food effect will be assessed in Part A (SAD) of this study.
  Interventions: Drug: TD-6450

INTERVENTIONS:
Drug: TD-6450
Drug: Placebo
  Arms: MAD TD-6450; SAD TD-6450

SUMMARY:
This study consists of two parts, Parts A and B. Part A is a single ascending dose (SAD) study in healthy subjects. Part B is a multiple ascending dose (MAD) study in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a female of non-childbearing potential or male, who is healthy, nonsmoking, and 18 to 60 years old, inclusive, at screening. Females are considered to be of non childbearing potential if they have had a hysterectomy or tubal ligation (documentation required) or are postmenopausal (amenorrheic for at least 2 years) with a follicle stimulating hormone (FSH) level >40 IU/L
* Subject has a body mass index 18 to 30 kg/m2, inclusive, and weighs at least 50 kg.

Exclusion Criteria:

* Subject has evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease.
* Subject has an estimated creatinine clearance of <90 mL/min at Screening or Day -1, calculated using the Cockcroft-Gault equation.
* Subject has participated in another clinical trial of an investigational drug (or medical device) within 60 days prior to Screening, or is currently participating in another trial of an investigational drug (or medical device).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Adverse events | 28 days max

SECONDARY OUTCOMES:
Cmax | 28 days max
  Pharmacokinetics
Tmax | 28 days max
  Pharmacokinetics
AUC | 28 days max
  Pharmacokinetics
T1/2 | 28 days max
  Pharmacokinetics
Food effect on AUC value | 15 days max
  Measure difference between fasted and fed doses

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- ICON Development Solutions, San Antonio, Texas, United States

REFERENCES:
- [Derived] Carucci M, Duez J, Tarning J, Garcia-Barbazan I, Fricot-Monsinjon A, Sissoko A, Dumas L, Gamallo P, Beher B, Amireault P, Dussiot M, Dao M, Hull MV, McNamara CW, Roussel C, Ndour PA, Sanz LM, Gamo FJ, Buffet P. Safe drugs with high potential to block malaria transmission revealed by a spleen-mimetic screening. Nat Commun. 2023 Apr 7;14(1):1951. doi: 10.1038/s41467-023-37359-2. PMID 37029122